CLINICAL TRIAL: NCT02598570
Title: An Open-Label, Single-Arm, Multicenter Phase 1 Study Evaluating the Safety and Pharmacokinetics of Duvelisib in Japanese Subjects With Relapsed or Refractory Lymphoma
Brief Title: Study Evaluating Duvelisib in Japanese Subjects With Relapsed or Refractory Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-460
Record Dates: First submitted 2015-10-21; First posted 2015-11-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Lymphoma
Keywords: Relapsed Lymphoma; Phosphoinositide 3-kinase (PI3K) Inhibitor; Duvelisib; Japanese; Refractory Lymphoma
MeSH Terms: conditions — Lymphoma; Hereditary Sensory and Autonomic Neuropathies | interventions — duvelisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- duvelisib (Experimental): Duvelisib will be administered orally as a fixed dose in 28-day cycles.
  Interventions: Drug: duvelisib

INTERVENTIONS:
Drug: duvelisib — Duvelisib will be administered orally as a fixed dose in 28-day cycles.
  Other Names: IPI-145; ABBV-954

SUMMARY:
This study seeks to evaluate the safety and pharmacokinetics of duvelisib in Japanese participants with relapsed or refractory lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoma (excluding lymphoblastic lymphoma)
* Progressed during, refractory to, intolerant of, or ineligible for established therapy, or has a disease for which there is no established therapy
* Eastern Cooperative Oncology Group (ECOG) performance status lower than or equal to 2
* Life expectancy of at least 3 months

Exclusion Criteria:

* Any prior treatment with a PI3K inhibitor or Bruton's tyrosine kinase (BTK) inhibitor
* Ongoing treatment with chronic immune-suppressants
* Overt CNS lymphoma
* Inadequate hepatic, bone marrow, or renal function
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months
* Venous thromboembolic event requiring anticoagulation
* Presence of active systemic infection within 72 hours of treatment
* Human immunodeficiency virus (HIV) infection
* Pregnant or lactating women

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting Treatment-emergent Adverse Events | Throughout the study for approximately 2 years
  The number of participants reporting treatment-emergent adverse events.
Maximum Observed Plasma Concentration (Cmax) of Duvelisib | Cycle 1 Day 1, 8, 15, and 22 and on Day 1 of Cycles 2 - 5
Time to Maximum Observed Concentration (Tmax) of Duvelisib | Cycle 1 Day 1, 8, 15, and 22 and on Day 1 of Cycles 2 - 5
Area Under the Plasma Concentration-time Curve (AUC) of Duvelisib | Cycle 1 Day 1, 8, 15, and 22 and on Day 1 of Cycles 2 - 5

SECONDARY OUTCOMES:
Overall Response Rate | Throughout the study for approximately 2 years
  Overall Response Rate is defined as the proportion of participants with a confirmed response of complete (CR) or partial response (PR) based on the revised International Working Group (IWG) criteria.
Overall Survival | Throughout the study for approximately 2 years
  Overall survival is defined as the duration in weeks from the date of the first dose of study treatment until the date of death.
Progression Free Survival | Throughout the study for approximately 2 years
  Progression free survival is defined as the time from the date of the first dose of study treatment to the first documentation of progressive disease (PD) or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Site Reference ID/Investigator# 141826, Aichi
  - Site Reference ID/Investigator# 141595, Fukuoka
  - Site Reference ID/Investigator# 141594, Tokyo